CLINICAL TRIAL: NCT01595204
Title: Olympia-MITO13-validation of a Laparoscopic Score to Predict the Chance of Optimal Cytoreduction in Advanced Ovarian Cancer Patients: an Open-label Prospective Multicentric-trial.
Brief Title: Validation of a Laparoscopic Score to Predict the Chance of Optimal Cytoreduction in Advanced Ovarian Cancer Patients
Acronym: MITO13
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Prof. Giovanni Scambia, Medical Doctor, Catholic University of the Sacred Heart
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P/758/CE/2009
Record Dates: First submitted 2012-05-08; First posted 2012-05-09 (Estimated); Last update posted 2012-05-22 (Estimated); Status verified 2012-05

CONDITIONS: Cancer of Ovary
Keywords: Cancer of Ovary, laparoscopy, operability , score.
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Laparoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Diagnostic Laparoscopy (Experimental): Laparoscopy will be performed in each case of clinical/radiological suspicious primary advanced ovarian/peritoneal cancer.
  Interventions: Procedure: Diagnostic laparoscopy

INTERVENTIONS:
Procedure: Diagnostic laparoscopy — Laparoscopy will be performed in each case of clinical/radiological suspicious primary advanced ovarian/peritoneal cancer.
  After the introduction of the trocar and the optic, pneumoperitoneum is induced and one or two ancillary trocars are inserted in the iliac fossae bilaterally or where it is possible. A careful complete abdominal and pelvic inspection is carried out in order to identify any possible cause of non optimal cytoreduction. All peritoneal surfaces and the gutters are closely examined and the liver is evaluated by rotating the laparoscope 360° through the umbilical port using grasping forceps as retractors. The small bowel loops and mesentery are evaluated by carefully folding back the various intestinal segments. The pelvis is explored after the bowel loops are retracted in the upper abdomen when possible. At the end of laparoscopy, a PI value is elaborated, based on table given to participant centers.

SUMMARY:
Prospective multicenter study that aims to evaluate the learning curve of a laparoscopic score to predict possibility of optimal cytoreduction in patients with ovarian / tubal / peritoneal advanced at the time of first surgery. The study consists of subjecting all patients with a clinical suspicion and / or radiological diagnostic laparoscopy (SLPs).

Laparoscopy should be described and recorded in electronic form. After the procedure each patient will have a Laparoscopic-evaluation-form filled up with a laparoscopic score (PI). The minimum number of cases to be enrolled is 10 patients, in a minimum time of 1 year. The data collected and the video should be sent to the Center Coordinator, who will determine the adequacy of the procedure and the accuracy of the score enrollment is completed for each center. All eligible subjects will be considered by intention-to-treat population (ITT). For this phase of the study, it is not necessary know the outcome of the surgical patient (RT) or if it was then subjected to exploratory laparotomy or less.

DETAILED DESCRIPTION:
Results from large but retrospective studies clearly demonstrated that RT after primary surgery is the most important prognostic factor in AOC patients. Subsequently, several studies have shown a complete cytoreduction (RT=0) is associated with a statistically significant longer survival rate than minimal residual disease (RT=1-2 cm). As a consequence, a maximal surgical effort is considered the main goal to pursue in these patients.

However, data from the literature have shown that a certain percentage of AOC patients, variable between 10 and 80%, are still considered inoperable at time of primary surgery, and they are submitted to an unnecessary xipho-pubic laparotomy. This approach, beside affecting QoL, can be related to some complications and delay in starting chemotherapy. This result can be related to a series of variables, including patient's performance status, philosophy of the centre and skillness of the surgeon. Finally, the anatomic diffusion of the disease is described as one of the most limiting factor to an optimal cytoreduction.

In order to preoperatively identify patients with unresectable tumors, which can be spared an unnecessary exploratory laparotomy, several approaches have been attempted, including CA 125 serum levels and CT-scan. However, the accuracy of those parameters has been unsatisfactory, and limited by the retrospective nature of the studies and the highly variable rates of optimal cytoreduction in different series.

Laparoscopy is well-known to offer a direct and magnified vision of the peritoneal cavity and a better view of the upper abdomen. It allows the pathological assessment of the disease without an open surgical procedure, with a shorter operating time and better results in terms of post-operative morbidity. We first demonstrated in a pilot study that laparoscopy alone is able to provide the same information regarding the chance of optimal cytoreduction (RT<= 1cm) than standard laparotomy in clinically AOC patients. Since then, other investigators have confirmed the role of laparoscopy in the evaluation of the possibility of achieving optimal residual disease in the same clinical subset.

However, one of the major criticism to these studies was represented by the surgeon subjectivity in evaluating optimal debulking in relation to surgical team and operating room performances. Consequently, on the basis of previous published papers, we set up a quantitative predictive model, which provides each patient with a score, taking into account several laparoscopically-assessed sites of disease to objectively predict the chance of achieving optimal cytoreduction. This model gives each parameter (omental cake, diaphragmatic carcinosis, peritoneal carcinosis, superficial liver metastases, stomach infiltration, bowel infiltration and mesenteric retraction) a value of 2 (see "Statistical considerations").

Finally, we undertook a study to validate the performance of the model in a larger prospective series of AOC patients. For each laparoscopic parameter we have discussed and agreed the characteristics able to define a positive evaluation, especially those identifying the critical areas of surgical resection. This study confirmed that with a PI cut-off > 8, the percentage of inappropriate "no exploration" is 0, while the percentage of unnecessary exploration equals to 40.5%. In conclusion the laparoscopic subjective ability to predict optimal cytoreduction was definitively turned into an objective score.

Moreover, the laparoscopic score (Fagotti's score) has been validated externally in a centre different from the one where it was developed [19,20], demonstrating that predictive qualities of PI remain unchanged even if applied on a different population centre, with own surgical background. This report suggests that the limit of subjectiveness, characterizing the evaluation of ovarian cancer spread, tend to a solution.

Study design Phase I

1. Patients with a clinical/radiological suspicious primary advanced ovarian/peritoneal cancer should undergo the following pre-operative staging examinations: haematological and chemical parameters, including CA 125 serum levels, thorax-abdomen-pelvis CT-scan.
2. If inclusion criteria will be satisfied, an informed consent has to be signed before any surgical procedure.
3. Patients will be then submitted to an open laparoscopy with at least one ancillary trocar to evaluate the seven parameters previously described, assigning each one a score to obtain a global predictive index. PI score is calculated based on. A video has to be registered.
4. Patients'characteristics, including histological diagnosis, should be reported in the enclosed summarizing schedule. On the other hand, no additional information regarding the following treatment of the patient, i.e. abandoned vs. upfront surgery, RT or follow up are required during the preliminary phase 1.
5. Send Laproscopic form, pre-operative documents and Video to the coordinating centre.

For preliminary phase 1, a minimum number of 10 patients has to be enrolled in one year. Time and number of cases can be increased to reach the established accuracy rate > 80%.

The fairness of the laparoscopic PI value obtained in each specific centre will be established through the revision of film material by the coordinating centre and the accuracy will be calculated after realizing 10 cases. The centres achieving an accuracy rate > 80% can enter in the second phase of the study. Other centres will require further cases until the achievement of the objective.

All enrolled patients who receive the expected treatment will be considered intention-to-treat-population (ITT).

Participation to preliminary Phase I of the study is a necessary but not sufficient pre-requisite to adhere to Phase II. A new approval from the Ethical Committee is needed to enter into the Phase II.

Centres can withdraw from the study in any time, but a written explanation is required.

Phase II Only centres participating to Phase I can enter into Phase II trial, after achieving an accuracy rate >75%. A new approval from the Ethical Committee is needed to enter into the Phase II.

1. Patients with a clinical/radiological suspicious primary advanced ovarian/peritoneal cancer should undergo the following pre-operative staging examinations: haematological and chemical parameters, including CA 125 serum levels, thorax-abdomen-pelvis CT-scan.
2. If inclusion criteria will be satisfied, an informed consent has to be signed before any surgical procedure (Appendix 1).
3. Patients will be then submitted to an open laparoscopy with at least one ancillary trocar to evaluate the seven parameters previously described, assigning each one a score to obtain a global predictive index. PI score is calculated based on Appendix 2. No videos need to be registered.
4. Patients'characteristics, including histological diagnosis, should be reported in the enclosed summarizing schedule (Appendix 3). In this case additional information regarding the following treatment of the patient, i.e. abandoned vs. upfront surgery, RT and site, type of surgical procedures needed to obtain optimal cytoreduction, and follow up data are required (Appendix 4).
5. Send Appendices 2 and 3 to the coordinating centre. For phase 2 study, a minimum number of 100 patients should be enrolled in two years, overall.

Results regarding the primary objective of the study can be obtained immediately after the enrolment of all the patients. Secondary objectives of the study need at least a minimum follow-up of 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Patients with a diagnosis suspect for advanced ovarian cancer (FIGO stage III-IV)
* Life expectancy of at least 4 weeks
* Performance Status ≤ 2
* Adequate respiratory, hepatic, cardiological, medullar and renal function (Creatinine Clearance > 60 mL/min according to Cockcroft's formula)
* Compliant patient with psychological ability to follow the study procedures

Exclusion Criteria:

* Pregnancy or nursing.
* Inadequate respiratory, hepatic, cardiological, medullar and renal function, that avoid safe surgery.
* Patients with cancer mass occupying the entire abdomen or infiltrating abdominal wall.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2010-03; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
a prospective and multicentric validation of the laparoscopic score (PI), developed at the Catholic University of the Sacred Hearth (UCSC), to predict surgical outcome in primary AOC patients | 2 years
  The primary objective of this study is to obtain a prospective and multicentric validation of the laparoscopic score (PI), developed at the Catholic University of the Sacred Hearth (UCSC), to predict surgical outcome in primary AOC patients. In particular, we want to identify the PI cut-off value, at which AOC patients can be reasonably considered not optimally resectable (RT< 1 cm) in an expert referring centre for AOC treatment, thus avoiding an unnecessary exploratory xipho-pubic laparotomy.

SECONDARY OUTCOMES:
Multicentric prospective validation of a laparoscopic PI in AOC patients | 2 years
progression Free Survival; Overall survival | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Anna Fagotti, MD PhD, Principal Investigator — Catholic University of Sacred Heart; Giovanni Scambia, MD, Principal Investigator — Catholic University of Sacred Heart; Francesco Fanfani, MD, Principal Investigator — Catholic University of Sacred Heart